CLINICAL TRIAL: NCT06201403
Title: Mechanical Properties of Peripheral and Accessory Respiratory Muscles in Chronic Obstructive Pulmonary Disease Patients
Status: Recruiting | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Other Study IDs: COPD&Myoton
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD Group: Patients diagnosed with COPD at Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital
  Interventions: Diagnostic Test: Determination of biomechanical properties of muscles
- Healthy Group: Healthy individuals without any chronic or acute disease
  Interventions: Diagnostic Test: Determination of biomechanical properties of muscles

INTERVENTIONS:
Diagnostic Test: Determination of biomechanical properties of muscles — All evaluations will be performed with a MyotonPRO (Myoton AS., Tallinn, Estonia) digital palpation device. The data of the cases to be evaluated and the patterns related to the measurements will be transferred to the device by establishing a computer connection. Measurements will be performed unilaterally. The measurement point of the subjects' unilateral muscles will first be marked with a pencil. The physiotherapist will hold the device vertically and apply downward pressure (18N) to the muscle body. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement.

SUMMARY:
The biomechanical properties of accessory respiratory muscles and peripheral muscles of COPD and healthy subjects will be measured and compared with the MyotonPro device.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with group C and D COPD according to GOLD staging
* Having been using the same medications for the last 4 weeks
* No additional comorbid diseases of the orthopedic, neurological or cardiac system

Exclusion Criteria:

* Presence of another respiratory system disease other than COPD
* Patients who have had an acute COPD exacerbation in the last 4 weeks
* Patients experiencing COPD exacerbations during the study protocol
* Presence of fatty tissue at the measurement points, which may impair the measurement quality.
* Have already participated in another clinical trial within the last 30 days that may affect the results of the study.

Inclusion Criteria for Healthy Cases

* Being over 18 years of age
* Not having any diagnosed chronic disease
* Not being a smoker

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD and healthy adults
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
M.Sternocleidomastoideus (SCM) myotonometric measurement | 107 millisecond
  To measure the tension of the SCM, participants will be asked to lie supine on the bed. The evaluator will mark the central point with a pencil on the line connecting the mastoid process and the clavicle bone and then take the measurement. The physiotherapist will hold the device vertically and apply downward pressure (18N) to the muscle body. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M. Trapezius myotonometric measurement | 107 millisecond
  Participants will be instructed to sit comfortably in a chair with back support, lean their hips against the back of the chair, and keep their pelvis stationary with their feet on the floor and their hands in their lap. The shoulders will be in a neutral position, the knee and hip joints will be flexed to 90 degrees, and the trunk will remain upright. The measurement point of the upper trapezius is the midpoint of the connection between C7 and the acromion. The physiotherapist will hold the device vertically and apply downward pressure (18N) to the muscle body. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M. Biceps brachii myotonometric measurement | 107 millisecond
  While the participants are in a supine position, measurements will be taken from the middle between the lateral acromion and the medial border of the cubital fossa. The physiotherapist will apply downward pressure (18N) to the muscle body by holding the device vertically. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M. Pectoralis Major (PM) myotonometric measurement | 107 millisecond
  To measure the muscular characteristics of the PM, participants will be asked to lie in a supine position with their hips neutrally positioned and their knees fully extended. The measurement point of PM is the intersection of the vertical line from the midpoint of the clavicle and the horizontal line from the axilla. The physiotherapist will hold the device vertically and apply downward pressure (18N) to the muscle body. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M. Rectus abdominis (RA) myotonometric measurement | 107 millisecond
  Participants will lie in a supine position, with bilateral legs hip-knee flexed, feet supported on the bed. The muscle tone of the RA muscle portion will be measured from a point approximately 3 cm next to the belly button. The probe will be placed perpendicular to the surface and pressure will be applied until the probe turns green. The physiotherapist will hold the device vertically and apply downward pressure (18N) to the muscle body. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M.Rectus femoris myotonometric measurement | 107 millisecond
  While the participants are in the supine position, measurements will be taken from the midpoint between the SIPS and the top of the patella. The physiotherapist will hold the device upright and apply downward pressure (18N) to the muscle body. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M.Vastus lateralis myotonometric measurement | 107 millisecond
  While the participants are in the supine position, measurement will be taken from the midpoint of the line from the upper pole of the patella to the greater trochanter. The physiotherapist will apply downward pressure (18N) to the muscle body by holding the device vertically. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement
M. Tibialis anterior myotonometric measurement | 107 millisecond
  While the participants are in the supine position, measurements will be taken from the head of the fibula to the medial malleolus and 2 cm laterally from one-third of the tibia. The physiotherapist will apply downward pressure (18N) to the muscle body by holding the device upright. When the red light on the plexiglass frame of the device probe turns green, the pressure application will be stopped and will remain constant until 5 strokes are made. In every 5 beats, the duration of 1 beat is 15 ms and the time between beats is 8 ms. The SENIAM sensor location guide will be considered as a reference for the estimated motor point determination in the MyotonPRO measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided